CLINICAL TRIAL: NCT04350060
Title: Memory Care of the Future: Improving the Quality of Dementia Care Through Innovative Redesign of the Memory Care Environment
Brief Title: Improving the Quality of Dementia Care Through Innovative Redesign of the Memory Care Environment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ying Ying (Christina) Chen, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-002202
Record Dates: First submitted 2019-12-18; First posted 2020-04-16 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Subjects with dementia will be living in a retro-fitted room with technological enhancements for a 12 month period.
  Interventions: Other: Retro-fitted room with technological enhancements
- Standard of Care Group (No Intervention)

INTERVENTIONS:
Other: Retro-fitted room with technological enhancements — Reconstructing and retrofitting a currently existing memory care room at Samaritan Bethany Arbor Terrace Senior Living with integrated technologies specifically to accommodate the needs of persons with dementia to enhance sensory stimulation in sight, sound and sleep.
  Arms: Intervention Group

SUMMARY:
Research study is being done to demonstrate novel opportunities to transform the way the dementia community is cared for.

ELIGIBILITY:
Inclusion Criteria:

* Patients currently residing at Arbor Terrace memory care unit
* Patients diagnosed with dementia

Exclusion Criteria:

* Hospice patients with less than 30 days of life expectancy at the time of enrollment

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-02-02 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2025-06-09 (Actual)

PRIMARY OUTCOMES:
Change in quality of life, as measured by the Quality of Life in Alzheimer's disease (QOL-AD) | every 2 weeks for up to one year
  Measured using the self-reported QOL-AD questionnaire comprised of 13 questions with a scale of poor = 1, fair = 2, good = 3, excellent =4. Scores range from 13 to 52, with higher scored indicating better quality of life.
Change in sleep quality, as measured by the Pittsburgh Sleep Quality Index (PSQI) | every 2 weeks for up to one year
  Measured using the self-reported PSQI that uses 9 questions regarding sleep quality to determine a final score where a total of "5" or greater is indicative of poor sleep quality.
Change in dementia related behaviors and delirium, as measured by the Neuropsychiatric Inventory-Questionnaire (NPI-Q) | every 2 weeks for up to one year
  Measured using the self-reported NPI-Q questionnaire that reports Yes = present or No = absent on 12 domains. If yes, then the informant rates the severity of the symptoms on a 3-point scale (1 = mild, 2 = moderate, 3 = severe) and the distress of the symptoms on a 5-point scale (0 = not distressing at all, 1 = minimal, 2 = mild, 3 = moderate, 4 = severe, 5 = extreme or very severe).
Change in mood, as measured by the Patient Health Questionnaire 9 (PHQ-9) | every 2 weeks for up to one year
  Measured using the self-reported PHQ-9 questionnaire that uses 9 question regarding patient health with a sale of not at all = 0, several days = 1, more than half the days = 2, nearly everyday =3. Scores range from 0 to 27, with higher scored indicating grater severity of depression.
Change in function and independence, as measured by the Katz Index of Independence in Activities of Daily living (KATZ) | every 2 weeks for up to one year
  Measured using the self-reported KATZ questionnaire with a scale of independence = 1 and dependence = 0 to determine total score. The KATZ ranges from 0 to 6 with the lower score indicated patient is very dependent and the higher score indicated patient is independent.
Change in medication use | every 2 weeks for up to one year
  Measured using recorded medication use from patient's chart.
Change in falls | monthly for up to one year
  Measured using recorded fall data from patient's chart.

SECONDARY OUTCOMES:
Change in caregiver burden, as measured by the Caregiver Strain Index (CSI) | 6 months
  Measured using the self-reported CSI questionnaire with a scale of Yes=1 and No=0. Total score of 7 or higher indicates a high level of stress.

OTHER OUTCOMES:
Change in emergency room and hospitalizations | monthly for up to one year
  Measured using recorded emergency room and hospitalization data from patient's chart.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Ying Chen, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No